CLINICAL TRIAL: NCT03880357
Title: Multi-center, Double-blind, Randomized, Placebo Controlled, Parallel-group Study Comparing Taro Product to RLD and Both Active Treatments to a Placebo Control in the Treatment of Scalp Psoriasis
Brief Title: To Evaluate the Therapeutic Equivalence and Safety in Treatment of Scalp Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTCS 1614
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Scalp Psoriasis
MeSH Terms: interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test Product (Experimental): Betamethasone Scalp Suspension 0.064%;0.0005% (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Betamethasone Scalp Suspension 0.064%;0.0005%
- Reference Product (Active Comparator): Taclonex® (Calcipotriene Hydrate and Betamethasone Dipropionate) Topical suspension 0.005%/0.064% (LEO PHARMA)
  Interventions: Drug: Taclonex®
- Placebo (Placebo Comparator): Vehicle of the test product (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Placebo topical suspension

INTERVENTIONS:
Drug: Betamethasone Scalp Suspension 0.064%;0.0005% — applied once daily by gently rubbing to the affected area(s) of the scalp for approximately 4 weeks.
  Other Names: Taclonex
  Arms: Test Product
Drug: Taclonex® — applied once daily by gently rubbing to the affected area(s) of the scalp for approximately 4 weeks.
  Other Names: Calcipotriene and Betamethasone Dipropionate
  Arms: Reference Product
Drug: Placebo topical suspension — applied once daily by gently rubbing to the affected area(s) of the scalp for approximately 4 weeks.
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
To demonstrate the superiority of the efficacy of the test and reference products over that of the placebo control in the treatment of scalp psoriasis.

DETAILED DESCRIPTION:
Multi-center, double-blind, randomized, placebo controlled, parallel-group study comparing test and reference products to a placebo control in the treatment of scalp psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female aged ≥18 years
* All male subjects had to agree to use accepted methods of birth control with their partners, from the day of the first application of the study drug to 30 days after the last application of the study drug
* Willing and able to understand and comply with the requirements of the protocol, including attendance at the required study visits
* A clinical diagnosis of stable (at least 6 months) scalp psoriasis involving at least 10% of the scalp

Exclusion Criteria:

* Female subjects who were pregnant, nursing, or planning to become pregnant during study participation
* Known hypersensitivity to calcipotriene, betamethasone dipropionate, other corticosteroids, or to any ingredients in the study drugs
* Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative, or pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
treatment success on the Physician's Global Assessment (PGA) of disease severity | Study Week 4 (Day 28 ± 4 days)
  The proportion of subjects in each treatment group with "treatment success" (defined as none or minimal, a score of 0 or 1, within the treatment area) on the PGA of disease severity
clinical success on the Physician's Global Assessment (PASI) of disease severity | Study Week 4 (Day 28 ± 4 days)
  The proportion of subjects in each treatment group with "clinical success" (defined as clear or almost clear, a score of 0 or 1, at the target lesion site) on the PASI. Each psoriatic sign of scaling, erythema and plaque elevation should have a score of 0 or 1 for the subject to be considered a clinical success. The target lesion is to be identified at Baseline as the most severe lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Yantovskiy, Study Director — Taro Pharmaceuticals
Locations (1):
- Catawba Research, LLC, Charlotte, North Carolina, United States